CLINICAL TRIAL: NCT04416152
Title: Impact of Female Pelvic Reconstruction Surgery on Lower Urinary Tract Symptoms, Psychosomatic Distress and Sexual Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital, Far Eastern Memorial Hospital
Other Study IDs: 109045-F
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No

INTERVENTIONS:
Procedure: Pelvic reconstruction surgery — Pelvic reconstruction surgeries, such as anterior/posterior colporrhaphy, sacrospinous ligament fixation, transvaginal mesh repair and sacrocolpopexy.

SUMMARY:
To get the impact of pelvic floor reconstruction surgery on lower urinary tract symptoms, psychological distress and sexual function.

ELIGIBILITY:
Inclusion Criteria:

* Women with pelvic organ prolapse, who will undergo pelvic reconstruction surgery
* Women who had undergone pelvic reconstruction surgeries in our hospital

Exclusion Criteria:

* Pregnant woman.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with pelvic organ prolapse, who will undergo or had undergo pelvic reconstruction surgeries.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-05-26 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the women's bladder function questionnaire of UDI-6 | 10 years
  Change of UDI-6 score between baseline and after pelvic reconstruction surgery. Score values 0-18, and higher scores mean a or worse outcome.
the women's bladder function questionnaire of IIQ-7 | 10 years
  Change of IIQ-7 score between baseline and after pelvic reconstruction surgery. Score values 0-18, and higher scores mean a or worse outcome.
Change of psychosomatic score | 1 year
  Change of psychosomatic score between baseline and after pelvic reconstruction surgery, and higher scores mean a or worse outcome.
Change of Overactive Bladder Symptom Score | 1 year
  Change of OABSS score between baseline and after pelvic reconstruction surgery. Score values 0-15, and higher scores mean a or worse outcome.
Change of FSFI score | 1 year
  Change of FSFI score between baseline and after pelvic reconstruction surgery. higher scores mean a or worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan